CLINICAL TRIAL: NCT04964570
Title: Digital Mental Health Care for COVID-19 High-Risk Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Director of PTSD team at Columbia University, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8128
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Stigma, Social; Help-Seeking Behavior
MeSH Terms: conditions — Social Stigma; Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video and behavioral change module (BCM) + booster (Experimental): Participants will watch the video and read the BCM twice (day 1 and day 14)
  Interventions: Behavioral: Video _ behavioral change module
- Video and behavioral change module (BCM) (Experimental): Participants will watch the video and read the BCM once (day 1 only)
  Interventions: Behavioral: Video _ behavioral change module
- Control (No Intervention): This arm will recieved the same length video with a content that is not related to mental health and no BCM

INTERVENTIONS:
Behavioral: Video _ behavioral change module — A short video (primary outcome) that aimed at reducing stigma towards treatments and increasing help seeking intentions.
  The behavioral change module (secondary outcome) is aimed at changing behaviors of sleep, exercise and social support.
  Arms: Video and behavioral change module (BCM); Video and behavioral change module (BCM) + booster

SUMMARY:
The mental health consequences of the COVID-19 pandemic are likely to be vast, exceeding the capacity of mental health services and delaying treatment for people in need, with devastating consequences for those affected. Emerging data suggest that frontline health workers (e.g. physicians, nurses, EMTs) and essential workers (in industries such as energy, and food products and services) face particular risks for mental health problems during and after the COVID-19 outbreak.

To address the unprecedented mental health needs during and as a result of the COVID-19 pandemic this study will develop and test novel, cost-effective and scalable, digitally-delivered mental health interventions, and will test this approach by focusing on health care workers and other essential workers.

DETAILED DESCRIPTION:
Stigma towards mental health care is a profound obstacle that interferes with individuals seeking these services. Research suggests that interventions that are based on social contact are the most efficient way to reduce stigma. By combining online video and interactive behavioral change modules, this study aims to address stigma and both empower essential workers (healthcare and non-healthcare workers) both to seek treatment for mental health issues as well as to reduce psychiatric symptoms by increasing social support, facilitating sleep hygiene, and maintaining physical exercise. A total of 4,200 members of these high-risk groups will be recruited to participate in a randomized controlled trial (RCT) testing the efficacy of the intervention.

The intervention will consist of brief videos in which empowered members of the respective high-risk group (presented by actors) share their COVID-19 related mental health problems and describe how they were able to confront their mental health problems, which in turn helped them seek mental health care. The video will be followed by a short, interactive, digital behavioral change module. Within each high-risk group, individuals will first be randomized to receive the video (one time), video plus booster (second administration of the video), or non-intervention video control.

The study will randomize participants within each high-risk group into one of three arms:

1) Video + Behavioral Change Module, with Booster: 2-3-minute video (in which empowered members of the respective high-risk group (protagonists) share their COVID-19 related mental health problems and describe how they were able to confront their mental health problems, which in turn helped them seek mental health care) will be followed by 3-4-minute online digital behavioral change modules at days 1 and 14 of the study ("video+booster"); 2) Video + Behavioral change modules without Booster: 2-3-minute video will be followed by 3-4-minute online digital behavioral change modules at day 1 only ("video"); 3) No Intervention video (Control Arm): Participants randomized to this arm will receive video not related to mental health ("control"). Following the intervention, the study includes three follow-ups (day 14, 30, and 90) to examine longer-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Essential workers (including healthcare workers)
* Age of 18-80
* US resident
* English speaker

Exclusion Criteria:

* N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4134 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Stigma (the SSOSH-3) | immediately after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Stigma (3 items of the SSOSH-3) | 14 days after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Stigma (3 items of the SSOSH-3) | 30 days after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Stigma (3 items of the SSOSH-3) | 90 days after the intervention
  Change in stigma items from baseline - higher score, indicate higher stigma (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) | Immediately after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) | 14 days after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) | 30 days after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)
Help Seeking Intentions (3 items of the ATSPPH) | 90 days after the intervention
  Change in treatment seeking intentions from baseline - higher score, indicate higher help seeking intentions (range of 3 to 12)

SECONDARY OUTCOMES:
Behaviors questionnaire | 14 days after the intervention
  Four questions about sleep (quality of sleep), exercise (amount of weekly exercise) and social habits (weekly number of people one contacted). We will measure change from baseline
Behaviors questionnaire | 30 days after the intervention
  Four questions about sleep (quality of sleep), exercise (amount of weekly exercise) and social habits (weekly number of people one contacted). We will measure change from baseline
Behaviors questionnaire | 90 days after the intervention
  Four questions about sleep (quality of sleep), exercise (amount of weekly exercise) and social habits (weekly number of people one contacted). We will measure change from baseline
Clinical outcome - Anxiety | 14 days after the intervention
  Change from baseline in GAD-7 (range 0-21, higher score indicate more anxiety)
Clinical outcome - Anxiety | 30 days after the intervention
  Change from baseline in GAD-7 (range 0-21, higher score indicate more anxiety)
Clinical outcome - Anxiety | 90 days after the intervention
  Change from baseline in GAD-7 (range 0-21, higher score indicate more anxiety)
Clinical outcome - Depression | 14 days after the intervention
  Change from baseline in PHQ-9 (range 0-27, higher score indicate more depression)
Clinical outcome - Depression | 30 days after the intervention
  Change from baseline in PHQ-9 (range 0-27, higher score indicate more depression)
Clinical outcome - Depression | 90 days after the intervention
  Change from baseline in PHQ-9 (range 0-27, higher score indicate more depression)
Clinical outcome - PTSD | 14 days after the intervention
  Change from baseline in PC-PTSD (range 0-5, higher than 2 indicates high probability of PTSD)
Clinical outcome - PTSD | 30 days after the intervention
  Change from baseline in PC-PTSD (range 0-5, higher than 2 indicates high probability of PTSD)
Clinical outcome - PTSD | 90 days after the intervention
  Change from baseline in PC-PTSD (range 0-5, higher than 2 indicates high probability of PTSD)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — NYSPI and Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No identifying data of participants will be shared

REFERENCES:
- [Derived] Amsalem D, Fisch CT, Wall M, Liu J, Lazarov A, Markowitz JC, LeBeau M, Hinds M, Thompson K, Smith TE, Lewis-Fernandez R, Dixon LB, Neria Y. The role of income and emotional engagement in the efficacy of a brief help-seeking video intervention for essential workers. J Psychiatr Res. 2024 May;173:232-238. doi: 10.1016/j.jpsychires.2024.03.027. Epub 2024 Mar 27. PMID 38554618
- [Derived] Amsalem D, Wall M, Lazarov A, Markowitz JC, Fisch CT, LeBeau M, Hinds M, Liu J, Fisher PW, Smith TE, Hankerson S, Lewis-Fernandez R, Neria Y, Dixon LB. Destigmatising mental health treatment and increasing openness to seeking treatment: randomised controlled trial of brief video interventions. BJPsych Open. 2022 Sep 16;8(5):e169. doi: 10.1192/bjo.2022.575. PMID 36111611
- [Derived] Amsalem D, Wall M, Lazarov A, Markowitz JC, Fisch CT, LeBeau M, Hinds M, Liu J, Fisher PW, Smith TE, Hankerson S, Lewis-Fernandez R, Dixon LB, Neria Y. Brief Video Intervention to Increase Treatment-Seeking Intention Among U.S. Health Care Workers: A Randomized Controlled Trial. Psychiatr Serv. 2023 Feb 1;74(2):119-126. doi: 10.1176/appi.ps.20220083. Epub 2022 Sep 13. PMID 36097721